CLINICAL TRIAL: NCT05121727
Title: Comparison of the Effects of Ultrasound-Guided Erector Spinae Plane Block and Combination of Deep and Superficial Serratus Anterior Plane Block on Postoperative Acute Pain in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Comparison of Erector Spinae Plane Block and Combination of Deep and Superficial Serratus Anterior Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-1862
Record Dates: First submitted 2021-10-23; First posted 2021-11-16 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pain, Postoperative; Thoracic Surgery, Video-Assisted; Erector Spinae Plane Block; Serratus Anterior Plane Block; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T5 spinous process, 20 ml of 0.25% bupivacaine hydrochloride will be injected into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: Erector Spinae Plane Block
- Deep and Superficial Serratus Anterior Plane Block (Active Comparator): In patients who are planned to have combined deep and superficial serratus anterior plane block, following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique beneath the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 10 ml 0.25% bupivacaine will be injected into the area. Then, with the same needle, will be returned 1-2 cm from the deep serratus anteror area to superficial serratus anteror area above the serratus anterior muscle and will be injected 2 ml normal saline for hydrodissection. Finally 10 ml of 0.25% bupivacaine will be injected for superficial serratus anetrior block into the interfacial area.
  Interventions: Procedure: Deep and Superficial Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, when the patient is placed in the lateral decubitus position. 20 ml of 0.25% bupivacaine will be used in applications.
  Arms: Erector Spinae Plane Block
Procedure: Deep and Superficial Serratus Anterior Plane Block — Combined Deep and Superficial Serratus Anterior Plane Block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, when the patient is placed in the lateral decubitus position. 20 ml of 0.25% bupivacaine will be used in applications.
  Arms: Deep and Superficial Serratus Anterior Plane Block

SUMMARY:
Video-assisted thoracic surgery (VATS) has become a common procedure in thoracic surgery. Severe postoperative pain may be encountered in patients undergoing VATS. Analgesic methods such as thoracic paravertebral block (TPVB), intercostal block and erector spina plane block (ESPB) are widely used for VATS. Among these methods, ultrasound (US) guided TPVB is the most preferred method. In recent years, the frequency of application of plane blocks as a component of multimodal analgesia has been increased. ESPB and SAPB are some of them. Generally, comparisons are made between ESPB and TPVB in studies and the analgesic effect is evaluated.There are two techniques for SAPB application. In Deep SAPB (DSAPB) application, local anesthetic agent is given under the serratus anterior muscle. In the Superficial SAPB (SSAPB) application, the local anesthetic agent is given above the serratus anterior muscle. Since it is done by entering from the same point in two applications, it is possible to perform these two applications at the same time with a single needle entry. The mechanisms of regional analgesia techniques used after thoracic surgery operations are also different from each other. Therefore, it may be possible to obtain a more effective analgesic effect in patients by combining the mechanism of action of DSAPB and SSAPB , as in the multimodal analgesia method. This study seeks to evaluate the effect of ESPB and combined DSAPB-SSAPB pain after VATS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-30 kg/m2
* Patients undergoing elective video assiste thoracoscopic surgery

Exclusion Criteria:

* Patient refusing the procedure
* History of chronic analgesic or opioid therapy
* History of local anesthetic allergy
* Infection in the intervention area
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | 1st, 2nd, 4th, 8th, 16th, 24th and 48th hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th, 24th and 48th hours after surgery.

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Postoperative intravenous morphine infusion therapy will be administered with patient-controlled analgesia (PCA) method. Thanks to PCA, how much morphine the patient needs will be followed in mg.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oostvogels L, Weibel S, Meissner M, Kranke P, Meyer-Friessem CH, Pogatzki-Zahn E, Schnabel A. Erector spinae plane block for postoperative pain. Cochrane Database Syst Rev. 2024 Feb 12;2(2):CD013763. doi: 10.1002/14651858.CD013763.pub3. PMID 38345071
- [Derived] Schnabel A, Weibel S, Pogatzki-Zahn E, Meyer-Friessem CH, Oostvogels L. Erector spinae plane block for postoperative pain. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013763. doi: 10.1002/14651858.CD013763.pub2. PMID 37811665